CLINICAL TRIAL: NCT04339842
Title: Eating Habits of Adults During the Quarantine
Status: Completed | Type: Observational
Sponsor: Eliz Arter (Other)
Collaborators: Kıbrıs İlim Üniversitesi (Other)
Responsible Party: Sponsor-Investigator, Eliz Arter, Sr. Instr., Eastern Mediterranean University
Organization: Eastern Mediterranean University (Other)
Other Study IDs: Nutr2020
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Health Behavior; Eating Behavior
Keywords: Coronavirus; Quarantine; Social Isolation; Eating Habits; Nutrition; COVID-19
MeSH Terms: conditions — Health Behavior; Feeding Behavior; Coronavirus Infections; Social Isolation; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults in quarantine due to the virus outbreak: Individuals over the age of 18 who spend most of their time at home in social isolation because of the Coronavirus to prevent the risk of contracting the virus
  Interventions: Other: Assessment of Dietary Changes in Adults in the Quarantine

INTERVENTIONS:
Other: Assessment of Dietary Changes in Adults in the Quarantine — The online survey will help to collect demographic data from the volunteers. Personal information and contact details, such as email, will not be asked. The survey will include questions about any increase or decrease in the consumption of main meals, snacks and fluid intake. If the participants of the study have observed changes in their dietary pattern since the beginning of the quarantine, details of these changes, such as an increase in the amount of main meal consumption, will be questioned.

SUMMARY:
The aim of this study is to assess the changes in the dietary habits of adults spending most of their time in their homes due to the Coronavirus (COVID-19) outbreak. Eating habits of individuals may vary greatly depending on several factors such as geographic location, socioeconomic conditions, education level, knowledge about nutrition and psychological factors. Since this period of quarantine is economically and psychologically stressful, we hypothesise that individuals may alter their usual eating habits.

DETAILED DESCRIPTION:
Since the World Health Organisation (WHO) declared the latest Coronavirus outbreak as a 'pandemic', most countries had to take strict measures such as travel bans and lock-downs to prevent the spread of the virus. Unfortunately, this unexpected situation has caused many people around to globe to panic buy and stock up on food for an unpredictable period of time as it cannot be estimated when the outbreak will be controlled.

Nutrition plays an important role in our everyday life; it makes up a large part of a healthy life, it brings individuals together to socialise around a table and sometimes it can be used in times of stress as a coping mechanism leading to emotional eating.

In this study it is hypothesised that adults may tempt to change their everyday eating habits due to social isolation. Humans are generally sociable beings and this period of social isolation will psychologically pressurise humans and may cause some of them to eat more in quantity or frequency as a mechanism to cope with the growing fear and anxiety. On the other hand, it is also hypothesised that, some individuals may prefer healthier ways of eating, such as consuming more fruits and vegetables, drinking more water etc, believing that if they can improve their immunity they will be less likely to contract the virus. The study may also show that some individuals will be highly impacted economically and this will alter their dietary preferences.

Within the scope of this study an online survey consisting of 20 questions will be asked to volunteers who are over the age of 18 and spend most of their time at home in social isolation because of the Coronavirus outbreak. The survey does not include any personal questions but only general demographic data including gender, age range, the country they are currently residing, quarantine duration and whether or not they have observed any changes in their eating patterns since the beginning of this period.

In some questions, observed changes, if any, are further investigated to include details such as increase/decrease in portion size, frequency of meals etc.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-80
* Spending most of their time at home in quarantine because of the Coronavirus outbreak not to contract the virus
* Having internet access
* Being able to read and comprehend English language

Exclusion Criteria:

* Having any mental impairment or degeneration
* Having any life-threatening health condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in Quarantine in their homes due to the COVID-19 outbreak
Sampling Method: Non-Probability Sample
Enrollment: 673 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in the Eating Habits of Adults during the Quarantine | One month
  This online survey will provide us with an idea of whether or not social isolation due to a pandemic will affect the usual eating patterns of adults either because of psychological stress or economic burden. It will also help us understand the context of these changes

CONTACTS AND LOCATIONS:
Overall Officials: Eliz Arter, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Online, Nicosia, Cyprus

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT04339842/Prot_SAP_000.pdf